CLINICAL TRIAL: NCT07360951
Title: THE EFFECTİVENESS OF OBSTETRİC VİOLENCE AWARENESS TRAİNİNG FOR MİDWİFERY STUDENTS: A ROLE-PLAYİNG-BASED APPROACH
Brief Title: ROLE-PLAYİNG BASED TRAİNİNG ON OBSTETRİC VİOLENCE AWARENESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Esra SABANCI BARANSEL, Assistant Professor, Inonu University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2024/6669
Record Dates: First submitted 2026-01-06; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Obstetric; Violence Against Women; Midwifery
Keywords: Role-playing,; Obstetric Violence; Awareness Training; Midwifery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental-Awareness group (Experimental): In the study, the Obstetric Violence Awareness Training Program (OVATP), structured around role-playing, was administered to students as group training by researcher. The OVATP program was completed in 8 sessions over 4 weeks for the students in the experimental group, with 2 sessions per day, once a week. To ensure active student participation, role-playing exercises were used in the sessions; scenarios involving obstetric violence and those consistent with a respectful birthing approach were dramatized. The role-playing activities were conducted with five third-year midwifery students from the same university. The scenarios were specially prepared by the researcher and finalized after obtaining the opinions of five experts working in the field. The scenarios were rehearsed by the researcher before implementation. The researcher manag
  Interventions: Behavioral: Obstetric Violence Awareness Training Program
- control (No Intervention): The control group received no training; the students continued with standard midwifery education processes.

INTERVENTIONS:
Behavioral: Obstetric Violence Awareness Training Program — The group that was not intervened
  Other Names: Control
  Arms: experimental-Awareness group

SUMMARY:
This study was conducted to determine the effects of obstetric violence awareness training given to midwifery students through the role-playing technique on the students' perception levels of obstetric violence and midwifery care behaviors.The study was conducted as a randomized controlled experimental study with 126 senior students (63 experimental, 63 control) studying midwifery at two public universities during the 2024-2025 academic year. Students in the experimental group received role-playing-based obstetric violence awareness training, while the control group received no intervention. Data were collected using the Student Personal Information Form, PercOV-S Q, and CBI-30. The effectiveness of the obstetric violence awareness training was assessed using pre-test and post-test measurements. Research hypotheses:

H1: Awareness training on preventing obstetric violence, delivered through role-playing techniques, enhances midwifery students' perceptions of obstetric violence.

H2: Awareness training on preventing obstetric violence, delivered through role-playing techniques, enhances midwifery students' perceptions of caring behaviors.

ELIGIBILITY:
Inclusion Criteria:• Being a final year midwifery student,

* Successfully completing the Pregnancy and Childbirth courses,
* Volunteering to participate in the research.

Exclusion Criteria:• Having previously received training on obstetric violence

* Having given birth before

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — women
Enrollment: 126 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Perception of Obstetric Violence in Students | 1 year
  The Perception of Obstetric Violence in Students Questionnaire (PercOV-S Q) was used to measure the perception levels of midwifery students regarding obstetric violence. This scale was developed by Mena-Tudela et al., and its adaptation into Turkish and a validity-reliability study were carried out by Yeniocak et al. A high total score on the scale indicates a high perception level of obstetric violence among students; a low score indicates a low perception level. The scale consists of 33 items and 2 subscales. These subscales were classified under two areas: "Protocolized-visible Obstetric Violence" and "Non-protocolized-invisible Obstetric Violence". The Cronbach's Alpha coefficient of the scale was determined to be 0.92.
Perception of Obstetric Violence in Students Questionnaire | 1 year
  The Perception of Obstetric Violence in Students Questionnaire (PercOV-S Q) was used to measure the perception levels of midwifery students regarding obstetric violence. This scale was developed by Mena-Tudela et al. and its adaptation into Turkish and a validity-reliability study were carried out by Yeniocak et al. A high total score on the scale indicates a high perception level of obstetric violence among students; a low score indicates a low perception level. The scale consists of 33 items and 2 subscales. These subscales were classified under two areas: "Protocolized-visible Obstetric Violence" and "Non-protocolized-invisible Obstetric Violence". The Cronbach's Alpha coefficient of the scale was determined to be 0.92.

SECONDARY OUTCOMES:
Caring Behaviors Inventory | 1 year
  The Caring Behaviors Inventory-30 (CBI-30) was used to measure students' perceptions of midwifery care. This scale was developed by Wolf et al, and its Turkish adaptation and validity-reliability study were conducted by Gül and Dinç. A high score on the scale indicates a high perception of midwifery care, while a low score indicates a low perception of midwifery care. The scale consists of 30 items and 3 subscales: "Respect for Others", "Professional Knowledge and Attitudes", and "Accessibility to the Individuals". The Cronbach's alpha coefficient of the scale was determined to be 0.97.

CONTACTS AND LOCATIONS:
Overall Officials: Kamile Esin TAŞDEMİR, Research Assistant, Principal Investigator — Amasya University; Esra SABANCI BARANSEL, Assistant Professor, Study Director — İnönü University
Locations (1):
- İnönü University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No patient